CLINICAL TRIAL: NCT04543032
Title: Effect of Sensorimotor Training on Gait, Ankle Muscle Strength and Quality of Life in Patients With Diabetic Peripheral Neuropathy: A Randomized Controlled Trial
Brief Title: Sensorimotor Training and Gait in Diabetic Polyneuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMT for polyneuropathy
Record Dates: First submitted 2020-08-31; First posted 2020-09-09 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): the patients in this group will receive sensorimotor training for 6 weeks in addition to medical care.
  Interventions: Other: sensorimotor training
- control group (No Intervention): the patients in this group will receive medical care only.

INTERVENTIONS:
Other: sensorimotor training — Sensorimotor exercises progressed from stable surfaces to unstable surfaces, training gait in a line (tandem walk or walking straight) followed by gait including change in directions, gait without obstacles to gait with obstacles, change in the support base (feet apart and then together), physical exercises with eyes opened and closed, always respecting the functional capacity of each patient and progressively increasing the difficulty of each exercise. To help the training, cones, balance board, bars, mats and a mini-trampoline will be used. According to the patient progress, the exercises will be combined, generating circuits
  Arms: study group

SUMMARY:
Diabetic peripheral neuropathy is a common chronic complication of diabetes mellitus which results in high public health costs and has a huge impact on patients' quality of life. It leads to sensory and motor deficits, which often result in mobility-related dysfunction, and alterations in gait characteristics. These alternations in gait performance cause increase in the risk of fall, which has the strongest association with symptoms of depression in patients with diabetes. However, little is known about possible treatment strategies for improving gait ability and reduce risk of fall in patients with diabetic neuropathy. So, the purpose of this study will be to investigate the effect of sensorimotor training on ankle muscle strength, gait and quality of life in patients with diabetic peripheral neuropathy.

To determine if there is an effect for sensorimotor training on gait, ankle muscle strength and quality of life in patients with diabetic peripheral neuropathy, the patient will be assessed before and after 6 weeks of treatment by measurement of ankle muscles strength using isokinetic dynamometer, measurement of different spatiotemporal gait parameters using gait trainer instrument , and assessment of quality of life of the patients using HRQL questionnaire (SF-36) before and after the treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* patient who have body mass index did not exceed 30 Kg/m2.
* type II diabetes mellitus diagnosed for at least 7 years.
* able to walk without assistance or assistive device
* able to stand on both feet and on one leg
* have controlled blood glucose level by the screening by Glycated Haemoglobin test (9 % > HbA1c > 6.5 %) .

Exclusion Criteria:

The patients will be excluded if they have:

* cognitive deficits, severe retinopathy, scares under their feet, hypo or hypertension, any medical conditions that would confound assessment of neuropathy such as malignancy, active/untreated thyroid disease, other neurological or orthopaedic impairments (such as stroke, poliomyelitis, rheumatoid arthritis, or severe osteoarthritis), and severe nephropathy that causes edema or needs haemodialysis.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Measurement of walking speed | change from baseline at six weeks
  Speed of walking is one of time variables for measurement of kinematic gait analysis. It measured by (meter/second).
  It will be measured using the Biodex Gait Trainer: It is a device designed specifically for assessment, rehabilitation and retraining of gait for all patients, which composed of a treadmill with an instrumented deck that monitors and records kinematic gait parameters with a high resolution color touch screen (Liquid-Crystal Display) attached to the treadmill to control the device settings and display results.
Measurement of step length | change from baseline at six weeks
  Step length is one of distance variables for measurement of kinematic gait analysis. It is the linear distance from the posterior aspect of the heel of one foot to the posterior aspect of the heel of the opposite foot and measured by (meter)
  It will be measured using the Biodex Gait Trainer
Measurement of stride length | change from baseline at six weeks
  Stride length is one of distance variables for measurement of kinematic gait analysis. It is the linear distance from the posterior aspect of the heel of one foot to the posterior aspect of the heel of the same foot and measured by (meter)
  It will be measured using the Biodex Gait Trainer

SECONDARY OUTCOMES:
Proprioception of ankle joint | change from baseline at six weeks
  proprioception of ankle joint will be measured by Biodex Isokinetic dynamometer system (Biodex Medical Incorporated., Shirley, New York, USA).
Muscle strength of ankle dorsiflexors and plantar flexors | change from baseline at six weeks
  The strength of the dorsiflexors and plantar flexors muscles of the ankle will be measured by Biodex Isokinetic dynamometer system (Biodex Medical Incorporated., Shirley, New York, USA).
Assessment of Quality of life | change from baseline at six weeks
  Quality of life will be measured by the Short-Form Health Survey (SF-36) questionnaire.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale.
  The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are:
  * vitality
  * physical functioning
  * bodily pain
  * general health perceptions
  * physical role functioning
  * emotional role functioning
  * social role functioning
  * mental health

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt

REFERENCES:
- [Background] Mkandla K, Myezwa H, Musenge E. The effects of progressive-resisted exercises on muscle strength and health-related quality of life in persons with HIV-related poly-neuropathy in Zimbabwe. AIDS Care. 2016;28(5):639-43. doi: 10.1080/09540121.2015.1125418. Epub 2016 Jan 5. PMID 26729347
- [Background] Monteiro RL, Sartor CD, Ferreira JSSP, Dantas MGB, Bus SA, Sacco ICN. Protocol for evaluating the effects of a foot-ankle therapeutic exercise program on daily activity, foot-ankle functionality, and biomechanics in people with diabetic polyneuropathy: a randomized controlled trial. BMC Musculoskelet Disord. 2018 Nov 14;19(1):400. doi: 10.1186/s12891-018-2323-0. PMID 30428863
- [Background] Mizukami H. [Pathophysiology of diabetic polyneuropathy]. Nihon Rinsho. 2016 Apr;74 Suppl 2:229-33. No abstract available. Japanese. PMID 27266093
- [Derived] Saleh MSM, Elbanna RHM, Abdelhakiem NM, Abdalla GAE. Sensorimotor Training Improves Gait, Ankle Joint Proprioception, and Quality of Life in Patients With Diabetic Peripheral Neuropathy: A Single-Blinded Randomized Controlled Trial. Am J Phys Med Rehabil. 2024 Jul 1;103(7):638-644. doi: 10.1097/PHM.0000000000002453. Epub 2024 Feb 29. PMID 38466203